CLINICAL TRIAL: NCT06487858
Title: A Multicenter Open-Label Phase 1a/1b Study to Evaluate the Safety and Preliminary Antitumor Activity of BGB-R046 as Monotherapy and in Combination With Tislelizumab in Participants With Selected Advanced or Metastatic Solid Tumors
Brief Title: A Study of BGB-R046 as Monotherapy and in Combination With Tislelizumab in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-R046-101
Record Dates: First submitted 2024-06-20; First posted 2024-07-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor
Keywords: BGB-R046; First-in-human; Advanced solid tumor; Anti-Programmed Death-1 (Anti-PD1)
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1a: Part A: Dose Escalation Monotherapy (Experimental): Sequential cohorts of increasing dose levels of BGB R046 will be evaluated as monotherapy.
  Interventions: Drug: BGB-R046
- Phase 1a: Part B: Dose Escalation Combination Therapy (Experimental): Sequential cohorts of increasing dose levels of BGB R046 will be evaluated in combination with tislelizumab.
  Interventions: Drug: BGB-R046; Drug: Tislelizumab
- Phase 1b: Dose Expansion and Dose Optimization (Experimental): The recommended dose(s) for expansion (RDFE) for BGB-R046 in combination with tislelizumab from Phase 1a will be evaluated in selected indications.
  Interventions: Drug: BGB-R046; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-R046 — Intravenous administration
Drug: Tislelizumab — Intravenous administration
  Arms: Phase 1a: Part B: Dose Escalation Combination Therapy; Phase 1b: Dose Expansion and Dose Optimization

SUMMARY:
This is a first-in-human (FIH) study that will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BGB-R046 as a single agent and in combination with tislelizumab (BGB-A317) in participants with advanced or metastatic immune-sensitive solid tumors.

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Participants able to provide a signed and dated written informed consent prior to any study-specific procedures, sampling, or data collection
* Participants with histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors who have previously received standard systemic therapy or for whom standard treatment is not available, not tolerated, or determined not appropriate based on the investigator's judgement
* ≥ 1 measurable lesion per RECIST v1.1
* Able to provide an archived tumor tissue sample
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Adequate organ function
* Life expectancy >12 weeks as determined by the investigator

Exclusion Criteria:

* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast)
* Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug(s)
* History of interstitial lung disease, noninfectious pneumonitis (including immune mediated), or uncontrolled lung diseases including pulmonary fibrosis, or acute lung diseases.
* Experienced ≥ Grade 3 imAE(s) on prior immuno-oncology agent (anti-PD-1, anti CTLA4, or other experimental drugs)
* Uncontrolled diabetes > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management, or ≥ Grade 3 hypoalbuminemia ≤ 14 days before the first dose of study drug(s).
* Infection (including tuberculosis infection, or other) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before the first dose of study drug(s)
* Immunodeficiency as assessed by the investigator to be not suitable for treatment with immune modulating anticancer agents

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participant with Adverse Events, Serious Adverse Events, Adverse Events of Clinical Interest and Dose-limiting Toxicities | Up to approximately 2 years
  Number of participants with AEs including serious adverse events (SAEs), defined as any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of study drugs, whether considered related to study drugs or not as graded by the National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI CTCAE) V5.0/American Society for Transplantation and Cellular Therapy (ASTCT) for cytokine release syndrome [CRS] and immune effector cell associated neurotoxicity syndrome [ICANS])
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-R046 | Up to approximately 2 years
  MTD is defined as the highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30% or the highest dose administered, respectively
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BGB-R046 | Up to approximately 2 years
  The potential RDFE[s] of BGB-R046 administered as monotherapy and in combination with tislelizumab will be determined based on the totality of the data and will also take in consideration the long term tolerability, pharmacokinetics, preliminary antitumor activity and any other relevant data available
Phase 1b: Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) as determined by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to approximately 2 years
  ORR is defined as the percentage of participants with confirmed CR or PR as determined by investigators per RECIST v1.1
Phase 1a: Time to Response (TTR) | Up to approximately 2 years
  TTR is defined as the time from the date of the first dose of study drug(s) to the date of the first determination of overall response by the investigator using RECIST v1.1
Phase 1a: Clinical Benefit Rate (CBR) | Up to approximately 2 years
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks
Phase 1a and Phase 1b: Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first objective response until the first documentation of disease progression after treatment initiation or death, whichever comes first, as determined by investigators per RECIST v1.1
Phase 1a and Phase 1b: Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants with the best overall response (BOR) of confirmed CR, PR, or stable disease, as determined by investigators per RECIST v1.1
Phase 1b: Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first administration of study drug to the date of the first documentation of disease progression or death due to any cause, whichever occurs first, as determined by investigators per RECIST v1.1
Phase 1b: Number of Participants with Adverse Events (AEs) | Up to approximately 2 years
  Number of participants with AEs, including serious adverse events (SAEs), defined as any unfavorable and unintended sign (including abnormal laboratory findings, physical examination, or electrocardiogram results), symptom, or disease temporally associated with the use of study drugs, whether considered related to study drugs or not as graded by NCI-CTCAE V5.0 or ASTCT as appropriate
Phase 1a: Plasma concentrations of BGB-R046 analytes | Predose and at select time points in Cycles 1, 2 and 5; predose at select Cycles between Cycles 3 and 25 (each cycle is 21 days); and at the first safety follow-up visit (conducted 30 days after the last dose of study drug)
Phase 1b: Plasma concentrations of BGB-R046 analytes | Predose and after end of infusion in Cycles 1 and 5; predose at select Cycles between Cycles 1 and 25 (each cycle is 21 days); and at the first safety follow-up visit (conducted 30 days after the last dose of study drug)
Phase 1b: Plasma concentrations of tislelizumab | Predose and after end of infusion in Cycles 1 and 5; predose at select Cycles between Cycles 1 and 17 (each cycle is 21 days); and at the first safety follow-up visit (conducted 30 days after the last dose of study drug)
Phase 1a and 1b: Maximum observed plasma concentration (Cmax) of BGB-R046 | Cycle 1 and Cycle 5 (each cycle is 21 days)
Phase 1a and 1b: Minimum Observed Plasma Concentration (Ctrough) Of BGB-R046 | Cycle 1 and Cycle 5 (each cycle is 21 days)
Phase 1a and 1b: Area Under the Plasma Concentration-time Curve (AUC) of BGB-R046 | Cycle 1 and Cycle 5 (each cycle is 21 days)
Phase 1a and 1b: Terminal Half-Life (t1/2) of BGB-R046 | Cycle 1 and Cycle 5 (each cycle is 21 days)
Phase 1a and 1b: Incidence of Antidrug Antibodies (ADAs) to BGB-R046 and tislelizumab | Periodic sampling up to Cycle 25 (each cycle is 21 days) and at the first safety follow up visit up to approximately 2 years (conducted 30 days after the last dose of study drug)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (8):
- China (8):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/